CLINICAL TRIAL: NCT05614908
Title: Nonsurgical Treatment of Achilles Tendon Rupture: Comparison of an 8-week Liberal Regime With an 11-week Restrictive Regime. A Prospective Cohort Quality Assurance Study.
Brief Title: Outcome After Conservatively Treated Achilles Tendon Rupture
Status: Enrolling by invitation | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Mette Frank Fenger, Principal Investigator, Aarhus University Hospital
Other Study IDs: AarhusUH-MFenger
Record Dates: First submitted 2022-11-03; First posted 2022-11-14 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Achilles Tendon Rupture; Achilles Tendon Injury
Keywords: Achilles tendon rupture; Functional ability; Immobilization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Achilles tendon rupture: Patients treated non-surgically at Aarhus University Hospital from 2022 to approximately 2028. Comparing an 8 week liberal regime wtih an 11 week restrictive regime.
  Interventions: Other: 11 week restrictive regime; Other: 8 week liberal regime

INTERVENTIONS:
Other: 11 week restrictive regime — As part of standard care at AUH (until May 2024), patients are immobilized in scotch cast with the foot in plantarflexion during week 0-4. Next, the scotch cast is replaced by a ROM-WALKER in plantarflexion for the next 7 weeks (week 5-11 after injury). The ROM-WALKER is gradually corrected from 30 degrees plantarflexion to 0 degrees. No weight bearing or exercises is allowed and they are not allowed to remove the ROM-WALKER during week 0-10. At week 11, the patients are allowed weight bearing up to 30 kg, after which there is no longer weight bearing restrictions.
  From week 12 they are allowed full weight bearing with a 1 cm heel lift i their shoes.
Other: 8 week liberal regime — The patients are treated with a walker orthosis with 3 wedges in plantarflexion, during week 1-2 with no weight bearing and no exercises. After 2 weeks, the tendon will be examined, and if no defect in the tendon is detected by palpation, the patients will start partially weight bearing in week 3-5, and full weight-bearing week 6-8. They are instructed in unloaded exercises for the calf and anklejoint after 2 weeks, and loaded exercises (elastic) after 5 weeks, with a maximum position til 0 degrees in the anklejoint. Balancetraining and stationary bike training after 7 weeks. The wedges are removed one by one after 3, 5 and 7 weeks, respectively.
  If there is a palpable defect in the tendon after 2 weeks, the patient must wait 1 week with partially weight bearing and exercises, and remove the wedges at 4, 5 and 7 weeks after the initiation of treatment.
  From week 9, walking i their shoes with a 1 cm heel lift.

SUMMARY:
The main purpose of the study is to compare the patient-reported outcomes and adverse events of two different rehabilitation regimes for patients undergoing non-surgical treatment of Achilles Tendon Rupture. Thus, using a pre-post study design we will compare whether patients participating in an 8-week liberal rehabilitation regime will achieve the same, or better, self- reported functional ability, without increased risk of adverse events, in the first two years following injury, compared to an 11 weeks more restrictive rehabilitation regime..

DETAILED DESCRIPTION:
Background:

The Achilles tendon is the most commonly injured tendon in the lower extremity, and can be treated either surgical or non-surgical. Previous studies have investigated early controlled motion and weight-bearing for non-surgically treated Achilles Tendon Rupture (ATR). Early motion may cause tendon elongation, which leads to decrease in push off strength, and thus potentially a poorer functional outcome. Conversely, delayed initiation of mobilisation and weight-bearing may similarly hinder or delay optimal recovery of function and return to work and sports. The correct treatment and rehabilitation, including the timing of rehabilitation initiation, may therefore be crucial to ensure the patients functional ability.

Most hospitals in Denmark treating patients with ATR, provide a regime of 8-9 weeks of treatment for non-surgically treated patients. At Aarhus University Hospital (AUH), however, a more restrictive regime has been provided for these patients in the past 7 years, with a treatment period of 11 weeks after injury, and with no or limited weight-bearing or exercises.

A previous retrospective study at AUH including 100 patients undergoing non-surgical treatment and the restrictive 11 week rehabilitation regime was conducted in 2023. The results documented a re-rupture rate of 4 %, comparable to the rate reported at the Danish ATR Database, and similarly comparable results on patient-reported disability measured with the Achilles tendon Total Rupture Score (ATRS). The Danish ATR Database includes data from 11 different hospitals in Denmark, where the majority have implemented a more liberal rehabilitation regime of 8-9 weeks of treatment with early weight-bearing and exercises. As a result of this retrospective study, we are changing the rehabilitation protocol of ATR at AUH, from 11 weeks restrictive regime, to an 8 weeks liberal regime.

Purpose:

With this quality assurance study we aim to compare patient-reported outcomes and adverse events in patients participating in an 8-week liberal regime compared to an 11-week restrictive regime following non-surgically treated ATR

Study design and setting:

This is an observational cohort study with prospectively collected patient-reported outcomes, conducted at AUH. First, 110 consecutive patients will be included while the existing 11-week restrictive regime is standard care, then the 8-week liberal regime will be implemented, and subsequently another 110 patients will be consecutively included.

Data collection procedures and outcomes:

Patients will receive a digital letter with a link to an online questionnaire to be completed at 6 months, 12 months and 24 months from the date of the treatment start.

Patients are asked to fill out the ATRS on functional ability, as well as additional questions regarding job status, return to sport, incidence of deep venous thrombosis, whether they have sustained a re-rupture, and their satisfaction with treatment they received at the hospital.

The ATRS is a 10-item questionnaire, with a score of 0 to 10 (worst-best), which has been found valid, reliable and responsive in this population.

Statistical analysis:

The primary outcome is the difference in the self-reported ATRS score at 12 months in patients participating in the 8-weeks regime compared to the 11-week regime.

The sample size needed to detect a minimal clinical important difference of 10 points (SD 18) between the two groups is 102, with a significance level of 5% and a power of 80%. To allow for subgroup analysis and with an estimated rate of drop-out of 20%, a minimum of 200 patients will be included.

ELIGIBILITY:
Inclusion criteria:

* Patients with an acute achilles tendon rupture treated non-surgically at AUH
* Treatment start maximum 14 days after time of rupture
* ≥18 years
* Understand and read Danish

Exclusion criteria:

* Patients who have not followed the regime at AUH (e.g. terminated use of the ROM- walker prematurely or similar)
* Bilateral ATR or rupture of the opposite in the treatmentperiod

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of approx. 220 consecutive acute achilles tendon rupture patients, treated non-surgically at Aarhus University Hospital from 2022 to approximately 2028.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Self-reported ATRS score at 12 months after injury | 12 months post-injury
  Achilles tendon Total Rupture Score (ATRS) is a self-reported questionnaire with 10 items, summing up to a score of 0-100 points, with 100 points reflecting no disability. The primary outcome will be ATRS score at 12 months, but data will also be collected at 6 and 24 months to describe any changes over time.

SECONDARY OUTCOMES:
Percentage of participants with re-rupture at 12 months | 12 months post-injury
  Self-reported re-rupture with consisting information in the medical record.
Percentage of participants who have returned to previous working status at 12 months | 12 months post-injury
  Self-reported return to previous work (if at working age)
Extend of participants who have returned to sports activities at 24 months | 24 months post-injury
  Self-reported return to sports activities, on a 0-10 scale (worst-best)

CONTACTS AND LOCATIONS:
Overall Officials: Nanna Rolving, Ph.d., Study Director — Aarhus University Hospital, Department of physiotherapy and occupational therapy; Per Gundtoft, Ph.d., Study Director — Aarhus University Hospital, Department of Orthopaedics
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No